CLINICAL TRIAL: NCT03726554
Title: Comprehensive Reverse Shoulder: Porous Augmented Glenoid Baseplate and Mini Humeral Tray Post-Market Clinical Follow-up Study
Brief Title: Post-Market Study of Comprehensive Reverse Augmented Glenoid and Mini Humeral Tray in Total Shoulder Arthroplasty
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMG2017-70E
Record Dates: First submitted 2018-09-26; First posted 2018-10-31 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Arthropathy of Shoulder Region; Grossly Deficient Rotator Cuff; Osteoarthritis of the Shoulder; Rheumatoid Arthritis Without Humeral Metaphyseal Defects; Post-Traumatic Arthritis
Keywords: Reverse Shoulder Arthroplasty; Medical Device; Performance; Safety; Shoulder Prosthesis; Glenoid Erosion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Comp. Rev. Porous Augmented Glenoid (Experimental): Subjects with a grossly deficient rotator cuff in need of a reverse shoulder arthroplasty who met the inclusion/exclusion criteria and received the Comprehensive Reverse Porous Augmented Glenoid.
  Interventions: Device: Comprehensive Reverse Porous Augmented Glenoid
- Comp. Rev. Mini Humeral Tray (Experimental): Subjects with a grossly deficient rotator cuff in need of a reverse shoulder arthroplasty who met the inclusion/exclusion criteria and received the Comprehensive Reverse Mini Humeral Tray
  Interventions: Device: Comprehensive Mini Humeral Tray

INTERVENTIONS:
Device: Comprehensive Reverse Porous Augmented Glenoid — Three glenoid baseplate options designed for various severities of glenoid erosion and deformity, the device promotes bony ingrowth while restoring natural human anatomy.
  Arms: Comp. Rev. Porous Augmented Glenoid
Device: Comprehensive Mini Humeral Tray — The mini humeral tray offers additional sizing options to the Comprehensive Shoulder line. The mini tray is designed to fit smaller anatomies.
  Arms: Comp. Rev. Mini Humeral Tray

SUMMARY:
This study is a multicenter, prospective, non-randomized, non-controlled, dual cohort post market surveillance study. The primary objective of this study is to confirm the safety and performance of the Comprehensive Reverse Shoulder System when used with the Comprehensive Porous Augmented Glenoid Baseplate and/or Comprehensive Mini Humeral Tray in primary and revision reverse shoulder arthroplasty.

DETAILED DESCRIPTION:
The Comprehensive Reverse Porous Augmented Glenoid Baseplate and Comprehensive Mini Humeral Tray belong to the Comprehensive Reverse Shoulder Arthroplasty System. They were developed to provide patients with grossly deficient rotator cuffs with another surgical option. The aim of the Comprehensive Reverse Shoulder System is to increase shoulder function while reducing pain.

A maximum of 7 sites will contribute to this study. Enrollment of 7 sites on a global scale will allow for assessment of device consistency across different regions. Enrollment per site will not exceed 45 shoulders. 146 implants will be included in this study with competitive enrollment. All potential study subjects will be required to participate in the Informed Consent process.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be 18 years of age or older.
* Patient must be anatomically and structurally suited to receive the implants and possess a functional deltoid.
* Patient must have a grossly deficient rotator cuff with severe arthropathy and/or a previously failed shoulder joint replacement with a grossly deficient rotator cuff.
* Patient must be able and willing to complete the protocol required follow-up.
* Patient must be able and willing to sign the Institutional Review Board/Ethics Committee approved informed consent.

Exclusion Criteria:

* Patient is a prisoner.
* Patient is a current alcohol or drug abuser.
* Uncooperative patient or patient with neurologic disorders who is incapable or unwilling to follow directions.
* Patient presents with osteoporosis.
* Patient has a metabolic disorder that may impair bone formation.
* Patient has osteomalacia.
* Patient has distant foci of infections which may spread to the implant site.
* Patient has rapid joint destruction, marked bone loss or bone resorption apparent on roentgenogram.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2018-08-28 (Actual); Primary Completion 2030-02 (Estimated); Study Completion 2030-02 (Estimated)

PRIMARY OUTCOMES:
Implant Survivorship | 10 years
  Based on removal or intended removal of the device and determined using the Kaplan-Meier method

SECONDARY OUTCOMES:
Frequency and Incidence of Adverse Events | 10 years
  Monitoring the frequency and incidence of adverse events, serious adverse events, adverse device effects, serious adverse device effects, and unanticipated serious adverse device effects as well as device deficiencies.
Clinical efficacy of the device is assessed using the American Shoulder and Elbow Surgeon Score Patient Questionnaire. | 10 years
  Pain, function, and activities of daily living are measured. The American Shoulder and Elbow Surgeon (ASES) scale is 0-100. 100 is the highest score and indicates the greatest function while 0 is the lowest score.
Radiographic Performance | 10 years
  X-rays will be evaluated for radiolucency, osteolysis, atrophy, hypertrophy, osteophytes, component migration, scapular notching and heterotopic ossification

CONTACTS AND LOCATIONS:
Overall Officials: Hillary Overholser, Study Director — Zimmer Biomet
Locations (6):
- United States (6):
  - Andrews Research and Education Foundation, Gulf Breeze, Florida
  - Norton Orthopedic Specialists, Louisville, Kentucky
  - William Beaumont Hospital, Royal Oak, Michigan
  - The Research Foundation for the State University of New York, Buffalo, New York
  - Campbell Foundation, Germantown, Tennessee
  - The Rector and Visitors of the University of Virginia, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No